CLINICAL TRIAL: NCT03791879
Title: The Analgesic Effectiveness and Safety of Upgraded Caudal Dexmedetomidine Doses in Pediatric Hypospadias Surgery.
Brief Title: Caudal Dexmedetomidine Analgesia in Pediatrics .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Latif Ghanim, Associate Professor os anesthesia ICU & Pain medicine., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MFM IR.18.11.322 - 2018/11/11
Record Dates: First submitted 2018-12-29; First posted 2019-01-03 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: 164 Boys for Hypospadias Surgery Under General Anesthesia With Caudal Block
Keywords: Caudal; Dexmedetomidine; Levobupivacaine; hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- • Group A will take Caudal Levob 0. 125%+ DEXM 0.5µg/k (Active Comparator)
  Interventions: Drug: Caudal dexamedatomidine analgesia
- • Group B will take Caudal Levob 0.125%+ DEXM 1µg/kg. (Active Comparator)
  Interventions: Drug: Caudal dexamedatomidine analgesia
- • Group C will take Caudal Levob 0. 125%+ DEXM 1.5 µg/ (Active Comparator)
  Interventions: Drug: Caudal dexamedatomidine analgesia
- • Group D will take Caudal Levob 0. 125%+ DEXM 2µg/kg. (Active Comparator)
  Interventions: Drug: Caudal dexamedatomidine analgesia

INTERVENTIONS:
Drug: Caudal dexamedatomidine analgesia — Technique performance (Caudal block): classical technique; palpation, identification and puncture with the patients in the lateral position (permits easy access to the airway under general anesthesia) using a 22-G short-beveled needle under sterile conditions advancing needle pierces the sacrococcygeal ligament.
  After needle insertion, pre-calculated volume of Levob plus DEXM bolus was injected as follow; Group A Caudal Levob 0.125%+ DEXM 0.5µg/kg. Group B Caudal Levob 0.125%+ DEXM 1µg/kg. Group C Caudal Levob 0.125%+ DEXM 1. 5 µg/kg. Group D Caudal Levob 0.125%+ DEXM 2µg/kg.

SUMMARY:
Dexmedetomidine (DEXM) is a highly selective α2-adrenoceptor agonist that has been used increasingly in pediatric anesthesia. This prospective double blinded randomized comparative study is designed to evaluate the analgesic effect of caudal increasing doses of DEXM 0.5 , 1 , 1.5 , 2µg/kg combined with Levobupivacaine (Levob) 0.125% (ED95% =125%=least effective concentration) in providing pain relief over a 24-h period and lowest surgical stress peak. Study hypothesis: Levobupivacaine 0.125 %( ED95) combined with different increasing doses of dexamedatomedine >1 µg/kg could not add more analgesic & stress response obtundation outcome, but increase side effects (sedation and hemodynamic depression). The peak cortisol level during urology surgery was at the end of the 1st postoperative (PO) hour. Aim of the Study: To detect the optimal analgesic and safe caudal adjuvant DEXM dose associated with the least side effects& stress response modulation, guided by PO Cortisol peak difference in between the study groups during pediatric hypospadias surgery.

DETAILED DESCRIPTION:
Background: Dexmedetomidine (DEXM) is a highly selective α2-adrenoceptor agonist that has been used increasingly in pediatric anesthesia. This prospective double blinded randomized comparative study is designed to evaluate the analgesic effect of caudal increasing doses of DEXM 0.5 , 1 , 1.5 , 2µg/kg combined with Levobupivacaine (Levob) 0.125% (ED95% =125%=least effective concentration) in providing pain relief over a 24-h period and lowest surgical stress peak. Study hypothesis: Levobupivacaine 0.125 %( ED95) combined with different increasing doses of dexamedatomedine >1 µg/kg could not add more analgesic & stress response obtundation outcome, but increase side effects (sedation and hemodynamic depression).The peak cortisol level during urology surgery was at the end of the 1st postoperative (PO) hour. Aim of the Study: To detect the optimal analgesic and safe caudal adjuvant DEXM dose associated with the least side effects& stress response modulation, guided by PO Cortisol peak difference in between the study groups during pediatric hypospadias surgery.

Optimal effective dose defined as; the least caudal DEXM dose which produce the best analgesic outcome [least time to 1st analgesic request and lowest rescue analgesic dose (24Hs)] associated with the least stress response (cortisol PO. first One hour peak), least PO sedation, and hemodynamic stability IO. &PO. HR & MAP. The peak cortisol level during urology surgery was at the end of the 1st postoperative (PO) hour.

. Material & Methods A prospective randomized double blinded (drug injector and PO assessor) comparative study will be conducted in Mansoura university hospital after obtaining ethics committee approval and written informed parental consent 164 boys (age 1-6 years, ASA I) scheduled for hypospadias surgery. Exclusion criteria; (Operative time exceeding 3 hours, bodyweight >25kg, bleeding diathesis, infection at the site of block, pre-existing neurological or spinal disease or abnormalities of the sacrum, inability to palpate the sacral hiatus by anatomic landmark palpation technique) or those with a history of allergic reactions to local anesthetics were excluded from the study. Patients will fast for solids 6h and water and 2 hours before surgery. After Patient Preoperative preparation, General anesthesia induction, caudal block and caudal drug injection (Levob plus DEXM) bolus will be injected according to each group as follow;

* Group A will take Caudal Levob 0. 125%+ DEXM 0.5µg/kg.
* Group B will take Caudal Levob 0.125%+ DEXM 1µg/kg.
* Group C will take Caudal Levob 0. 125%+ DEXM 1.5 µg/kg.
* Group D will take Caudal Levob 0. 125%+ DEXM 2µg/kg.

The study outcomes recording:

1ry outcome: Time to (1st analgesic request OPS >4). Secondary outcome: Total 24hours PO. Rescue analgesic dose IM pethidine 0.5mg/kg [2,3] based on local policy and protocol, Patients demographic data [age, weight, end tidal Sevoflurane (volume %) prior starting skin closure, intraoperative fentanyl total dose, recovery time (time from discontinuation of anesthesia to spontaneous eye opening)], Serum Cortisol level at basal before anesthesia and 1hour postoperative in between groups [1] , Apnea incidence (NO&%), and desaturation (NO&%), Objective pain score, Sedation score, Behavioral score for Agitation assessment, and Modified bromage score (residual Lower limb muscle weakness) recorded every 15 minutes for 1st hour then every 30 minutes for next 3 PO hours then at next 6th, 12th, 18th, 24th PO hours, hemodynamics, HR&SBP the incidence of bradycardia and hypotension per 50% percentile. Recorded every 10 minutes IO for maximum operative time 3 hours and every 30 min PO for next 2h in the recovery room until the child was discharged to the ward.

ELIGIBILITY:
Inclusion Criteria:

* 164 boys (age 1-8 years, ASA I) scheduled for hypospadias surgery

Exclusion Criteria:

* Operative time exceeding 3 hours, bodyweight >25kg, bleeding diathesis, infection at the site of block, pre-existing neurological or spinal disease or abnormalities of the sacrum, inability to palpate the sacral hiatus by anatomic landmark palpation technique) or those with a history of allergic reactions to local anesthetics were excluded from the study

Ages: 1 Year to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 164 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Time to (1st analgesic request objective pain score (OPS) ≥4) | Basal (0) till 24 hours.
  time from full recovery till child express moderate pain OPS 4 and ask for the first analgesic dose

CONTACTS AND LOCATIONS:
Overall Officials: mohamed A Ghanem, A professor, Study Chair — Mansoura Univeristy
Locations (1):
- Anesthesia department,Faculty of medicine, Mansoura univerisety, Al Mansurah, Egypt